CLINICAL TRIAL: NCT05185258
Title: An Investigator-Initiated, Phase 4, Open-Label, Single-Arm, Single-Center Study Investigating the Residual Disease Memory in Psoriasis Skin During Enstilar® and Narrow-Band Ultraviolet B Therapy: The Mempsolar Study
Brief Title: Residual Disease MEMory in PSOriasis Skin During EnstiLAR® and Narrow-band Ultraviolet B Therapy: The MEMPSOLAR Study
Acronym: MEMPSOLAR
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Thomas Emmanuel, Principal Investigator, Aarhus University Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: MEMPSOLAR
Record Dates: First submitted 2021-11-01; First posted 2022-01-11 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Psoriasis Vulgaris; Psoriasis; Skin Diseases; Skin Diseases, Papulosquamous; Skin and Connective Tissue Diseases
Keywords: Psoriasis; Narrowband UVB; NBUVB; T cell; T cells; Tissue-resident memory T cell; Tissue-resident memory T cells; Dendritic cells; Macrophages; Keratinocytes; Digital Spatial Profiling; GeoMX; NanoString; Regulatory T cells; Regulatory T cell; PASI; Immunohistochemistry; CD103; CD69; CD49a; Transcriptomics; TRM; Spatial; CD163; Topical; Foam; Calcipotriol/Betamethasone; Cal/Bet; Phototherapy; Disease Memory; Molecular Scar
MeSH Terms: conditions — Psoriasis; Skin Diseases; Skin Diseases, Papulosquamous; Skin and Connective Tissue Diseases | interventions — betamethasone dipropionate, calcipotriol drug combination

STUDY DESIGN:
Intervention Model Description: MEMPSOLAR is a phase 4, single-center, open-label, single-arm, self-controlled, split-body, interventional, vehicle-controlled, prospective cohort study evaluating the efficacy of Enstilar® foam in combination with NB-UVB in changing the number and/or type of TRM-cells in the skin in participants with moderate to severe psoriasis.
Masking Description: As no blinding or randomization is instituted the investigator and sponsor will know the patient number and treatment. Some aspects of the analysis will be performed blinded were possible.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Enstilar (Experimental): Participants will need to have two separate clinically healed psoriasis plaques. At baseline (visit 2), one target lesion (plaque # 1) will be actively treated with once-daily cutaneous application of Enstilar® foam and one target lesion (plaque # 2) will be treated with placebo-vehicle. Participants will then simultaneously be treated three-weekly with full-body NB-UVB for 8 weeks (or a minimum of 20 sessions in total). After 4 weeks of Enstilar® and emollient, treatment application will be changed to twice-weekly until EOT (visit 5). First dose of IMP will be administered by trained personal. Subsequent doses will be administered by the participant. Study visits will occur at Screening, Baseline (Week 0), Weeks 8, 13, and 18. At baseline, week 8, week 13, and week 18 two skin punch biopsies will be acquired from each target lesion.
  Interventions: Drug: Enstilar
- Placebo-vehicle (Placebo Comparator): Placebo-vehicle will be given as explained for the arm description under Enstilar.
  Interventions: Drug: Placebo-vehicle

INTERVENTIONS:
Drug: Enstilar — Topical foam
  Arms: Enstilar
Drug: Placebo-vehicle — Topical foam
  Arms: Placebo-vehicle

SUMMARY:
Psoriasis is a non-communicable chronic immune-mediated disease. Psoriatic skin is characterized by excessive proliferation of skin cells and infiltration of immune cells. The cause of psoriasis is so far unknown.

Established therapeutics include topical, oral-systemic, biologic, narrow-band ultraviolet B (NB-UVB). A persistent antipsoriatic effect by the newest biologic therapies has been demonstrated after treatment discontinuation. However, the remittive hallmark of psoriasis suggests the existence of a molecular scar, a kind of disease memory, in clinically healed skin. It has been suggested that this disease memory can be attributed to the tissue-resident memory T (TRM) cell.

The main purpose of the study is to investigate whether (NB-UVB) treatment and concomitant Enstilar® treatment can change the amount of TRMs in the skin as well as change the expression in the microenvironment around these cells in the skin from psoriasis patients. In addition, the investigators will investigate whether the treatment can change the quantity and types of other psoriasis-related cells in the skin. In addition to this, the investigators will also examine the effect of treatment on patient-related parameters.

ELIGIBILITY:
Inclusion Criteria:

Age:

1. Women or men with chronic stable plaque psoriasis aged 18 years or older at the time of consent. Consent must be obtained prior to any study-related procedures. The participants must furthermore be willing to participate and must be of a condition capable of giving informed consent.

   Type of participant and disease characteristics:
2. History of chronic stable plaque psoriasis.
3. Candidate for topical treatment, as judged by the investigator.
4. Candidate for NB-UVB treatment, as judged by the investigator.
5. Two target lesions of ~3 cm at its longest axis located on the body (except for the scalp, face, or intertriginous areas), scoring at least 1 for each of redness, thickness, and scaliness on the TPSS.
6. Women involved in any sexual intercourse that could lead to pregnancy must agree to use an effective contraceptive method from at least 4 weeks before baseline (visit 2). Effective contraceptive methods are: Systemic hormonal contraceptives (oral contraceptive, transdermal patches, vaginal rings, long-acting injectables, or implants), intrauterine devices, vasectomy, or barrier methods of contraception in conjunction with spermicide. This must be used until EOT. Hormonal contraceptives must be on a stable dose for at least 4 weeks before baseline (visit 2).

   a. Women of nonchildbearing potential are as follows: i. Women ≥60 years of age. ii. Women who have had surgical sterilization (hysterectomy, bilateral oophorectomy, bilateral salpingectomy, or bilateral tubal ligation) iii. Women >40 and <60 years of age who have had a cessation of menses for at least 12 months and a follicle-stimulating hormone (FSH) test confirming nonchildbearing potential (FSH ≥40 mIU/mL) or cessation of menses for at least 24 months without FSH levels confirmed.
7. A negative serum pregnancy test at screening and a negative urine pregnancy test at baseline (visit 2) must be presented by women of childbearing potential.

   Exclusion Criteria:

   Type of participant and disease characteristics:
8. Female participant who is breastfeeding, pregnant, or who is planning pregnancy during the study period.
9. History of concomitant skin disease or presence of skin condition that, in the opinion of the investigator, would interfere with the study assessments and the acquisition of biopsies.
10. Other psoriasis subtype (erythrodermic, guttate, pustular, inverse, drug-induced).
11. History or presence of signs or symptom of progressive or uncontrollable infectious, endocrine, neurological, renal, hepatic, cardiac, hepatic, vascular, pulmonary, gastrointestinal, hematological rheumatological, psychiatric or metabolic disturbance and/or abnormal blood test or vital signs other paraclinical information, including disorders of calcium metabolism, that, in the opinion of the investigator, may expose the patient to elevated or unnecessary risk or interfere with the interpretation of results.
12. Known hypersensitivity to any ingredient in the IMP or to components of the container.
13. Infectious skin lesions on treated areas (e.g., herpes, varicella, fungal, bacterial, and parasitic skin infections, skin manifestations in relation to tuberculosis).
14. Treated skin must not be affected by perioral dermatitis, striae atrophicae, atrophic skin, fragility of skin veins, ichthyosis, acne vulgaris, acne rosacea, rosacea, ulcers, and wounds.
15. History or presence of signs or symptoms of a light dermatosis (e.g., polymorphic light eruption, juvenile spring eruption, actinic folliculitis, actinic prurigo, solar urticaria, or chronic actinic/photosensitivity dermatitis.
16. Participant has had, or is planning, a major surgery within 8 weeks prior to baseline during the study.
17. Participant has a contraindication to skin biopsies.
18. Are taking medication known to cause phototoxic reactions (e.g., nonsteroidal anti-inflammatory drugs, tetracyclines, or thiazides).
19. Participant is currently receiving an investigational product or device or has received one within 4 weeks prior to baseline, that in the opinion of the investigator, might interfere with the results.
20. Participant has used biologic medication 12 weeks prior to baseline visit (Day 0), or 5 half-lives (whichever is longer).
21. Use of any systemic treatment for psoriasis (such as methotrexate, immunosuppressive drugs, corticosteroids, azathioprine, or cyclosporine) within 4 weeks prior to baseline.
22. Use of any topical medication to treat psoriasis (including salicylic acid, retinoid, calcineurin inhibitors, corticosteroids, vitamin D analogue, or tar) within 2 weeks prior to baseline. Use of moisturizers and emollients are not exclusion criteria.
23. Participant had psoralen and ultraviolet A (PUVA) treatment within 12 weeks prior to baseline.
24. Participant had any UVB phototherapy (including tanning beds) or excimer laser within 12 weeks prior to baseline.
25. Participant had excessive sun exposure within 2 weeks prior to baseline. This includes unwillingness to minimize natural and artificial sun exposure. Sunscreen products and protective apparel are recommended for circumstances when exposure cannot be avoided. Sunscreen must not be applied on the clinic visit days before the visit.
26. Participant has a history of an allergic reaction or significant sensitivity to lidocaine or other local anesthetics.
27. History of keloid formation or hypertrophic scarring in suture sites or scars.
28. Known inability or unavailability of a participant to complete required study visits during study participation.
29. A psychiatric condition (e.g., suicidal ideation) or chronic alcohol or drug abuse problem, determined from the participant's medical history, which, in the opinion of the investigator, may obstruct compliance.
30. Participant protected by the law (adult under guardianship, or hospitalized in a public or private institution for a reason other than study, or incarcerated).
31. Mental or linguistic incapacity to sign the consent form.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2022-02-16 (Actual); Primary Completion 2024-01-15 (Actual); Study Completion 2026-07-15 (Estimated)

PRIMARY OUTCOMES:
Evaluate the efficacy of Enstilar® foam in combination with NB-UVB in changing the TRM-cell number in the skin. | Up to 18 weeks
  Change in number of TRM-cells in the epidermis and dermis between baseline, week 8, week 13, and week 18.
  The following markers in combination will be used to differentiate cells: CD3, CD4, CD8, CD69, CD103.
Evaluate the efficacy of Enstilar® foam in combination with NB-UVB in changing the TRM-cell microenvironment in the skin. | Up to 18 weeks
  Change in the microenvironment surrounding TRM-cells in the epidermis between baseline, week 8, week 13, and week 18.
  The following markers in combination will be used to differentiate cells: CD3, CD4, CD8, CD69, CD103.

SECONDARY OUTCOMES:
Evaluate the efficacy of Enstilar® foam in combination with NB-UVB in changing CD11c+ cells using quantitative immunohistochemistry analysis over the study duration. | Up to 18 weeks
  Change in CD11c+ Dendritic cells.
  All assessments will be made between baseline, week 8, week 13, and week 18.
  Assessments will be reported as either/or: Counts/epidermal length, counts/area, positive stained area /epidermal length, or positive stained area/ area.
Evaluate the efficacy of Enstilar® foam in combination with NB-UVB in changing CD163+ cells using quantitative immunohistochemistry analysis over the study duration. | Up to 18 weeks
  Change in CD163+ Macrophages.
  All assessments will be made between baseline, week 8, week 13, and week 18.
  Assessments will be reported as either/or: Counts/epidermal length, counts/area, positive stained area /epidermal length, or positive stained area/ area.
Evaluate the efficacy of Enstilar® foam in combination with NB-UVB in changing Langerin+/CD207+ cells using quantitative immunohistochemistry analysis over the study duration. | Up to 18 weeks
  Change in Langerin+/CD207+ Langerhans-cells.
  All assessments will be made between baseline, week 8, week 13, and week 18.
  Assessments will be reported as either/or: Counts/epidermal length, counts/area, positive stained area /epidermal length, or positive stained area/ area.
Evaluate the efficacy of Enstilar® foam in combination with NB-UVB in changing Change in Myeloperoxidase+ cells using quantitative immunohistochemistry analysis over the study duration. | Up to 18 weeks
  Change in Myeloperoxidase+ cells
  All assessments will be made between baseline, week 8, week 13, and week 18.
  Assessments will be reported as either/or: Counts/epidermal length, counts/area, positive stained area /epidermal length, or positive stained area/ area.
Evaluate the efficacy of Enstilar® foam in combination with NB-UVB in changing FOXP3+ cells using quantitative immunohistochemistry analysis over the study duration. | Up to 18 weeks
  Change in FOXP3+ cells.
  All assessments will be made between baseline, week 8, week 13, and week 18.
  Assessments will be reported as either/or: Counts/epidermal length, counts/area, positive stained area /epidermal length, or positive stained area/ area.
Evaluate the efficacy of Enstilar® foam in combination with NB-UVB in changing Ki67+ cells using quantitative immunohistochemistry analysis over the study duration. | Up to 18 weeks
  Change in Ki67+ cells (also termed proliferation).
  All assessments will be made between baseline, week 8, week 13, and week 18.
  Assessments will be reported as either/or: Counts/epidermal length, counts/area, positive stained area /epidermal length, or positive stained area/ area.
Evaluate the efficacy of Enstilar® foam in combination with NB-UVB in changing CD49a+ cells using quantitative immunohistochemistry analysis over the study duration. | Up to 18 weeks
  Change in CD49a+ cells.
  All assessments will be made between baseline, week 8, week 13, and week 18.
  Assessments will be reported as either/or: Counts/epidermal length, counts/area, positive stained area /epidermal length, or positive stained area/ area.
Evaluate the efficacy of Enstilar® foam in combination with NB-UVB in changing the epidermal thickness over the study duration. | Up to 18 weeks
  • Change in epidermal thickness.
  The assessments will be made between baseline, week 8, week 13, and week 18. The epidermal thickness will be reported as epidermal area/epidermal length.
Evaluate the efficacy of Enstilar® foam in combination with NB-UVB in the whole transcriptome. | Up to 18 weeks
  Change in differentially expressed genes between baseline, week 8, week 13, and week 18.
Evaluate the efficacy of Enstilar® foam in combination with NB-UVB on changing the Psoriasis Area and Severity Index. | Baseline, Week 8, Week 13, Week 18
  Change between baseline, week 8, week 13, and week 18 for Psoriasis Area and Severity Index (PASI). PASI is the most widely used tool for assessing psoriasis severity in clinical trials. PASI is calculated as a measure of the average redness, thickness, and scaliness of the lesions (each graded on a 0-4 scale, with 0 being none and 4 being maximum), weighted by the involved body surface area in percentage. Results range from 0 to 72 with 0 being no disease and 72 being complete skin coverage with 4 in redness, 4 in thickness, and 4 in scaliness. Treatment response is assessed as PASI reduction in percentage. Every effort should be made to ensure that assessments will be performed by the same investigator at all visits including screening.
Evaluate the efficacy of Enstilar® foam in combination with NB-UVB on changing the 5-point Investigator's Global Assessment. | Baseline, Week 8, Week 13, Week 18
  Change between baseline, week 8, week 13, and week 18 for the 5-point Investigator's Global Assessment (IGA). The IGA is a static psoriasis severity assessment tool consisting of a 5-point ordinal scale ranging from ''clear'' to ''severe''. Every effort should be made to ensure that assessments will be performed by the same investigator at all visits including screening.
Evaluate the efficacy of Enstilar® foam in combination with NB-UVB on changing the Target Plaque Severity Score. | Baseline, Week 8, Week 13, Week 18
  Change between baseline, week 8, week 13, and week 18 for the Target Plaque Severity Score (TPSS). The TPSS is used in this study to bilaterally compare the treatment effect in localized psoriasis target plaques. The TPSS includes a measure of the redness, thickness, and scaliness of the lesion and is graded on a 0 to 4 scale (0 = clear, 1 = slight, 2 = mild, 3 = moderate, 4 = severe). The scores will be summed to produce the TPSS sum score. Furthermore, standardized target lesion images and subsequent computerized image analysis will be used to calculate the Target Plaque Area (TPA). Every effort should be made to ensure that assessments will be performed by the same investigator at all visits including screening.
Evaluate the efficacy of Enstilar® foam in combination with NB-UVB on changing the Dermatology Life Quality Index | Up to 18 weeks
  Change between baseline, week 8, week 13, and week 18 for the Dermatology Life Quality Index (DLQI). The DLQI is one of the most used validated questionnaires to assess the quality of life (QoL) associated with dermatological conditions. 10 items address the participant's perception of the impact of their skin disease on different aspects of their quality of life (QoL). Each item is scored on a 4-point Likert scale (0 = not at all/not relevant; 1 = a little, 2 = a lot, 3 = very much). The total score is the sum of the 10 items (0 to 30). A high score is indicative of a poor QoL. A 4-point change in the DLQI total score is normally referred to as a within-participant minimal important difference. A DLQI total absolute score of 0 or 1 indicates no or small impact of the disease on health related quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Emmanuel, M.D., Principal Investigator — University of Aarhus
Locations (1):
- Department of Dermatology, Aarhus N, Central Jutland, Denmark